CLINICAL TRIAL: NCT03319017
Title: The Impact of Hypoxic Conditions on Apoptosis in Polymorphonuclear Cells and Inflammatory Cytokines of Trauma Patients at Emergency Department
Brief Title: Apoptosis in Polymorphonuclear Cells and Inflammatory Cytokines of Trauma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Korea University (Other)
Responsible Party: Principal Investigator, Jung-Youn Kim, Assistant Professor, Korea University Guro Hospital
Other Study IDs: KUGH17229 (trauma)
Record Dates: First submitted 2017-10-17; First posted 2017-10-24 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Trauma
Keywords: Hypoxia; Hyperinflammatory; Hyperoxia; Apoptosis; Oxygenation; Polymorphonuclear Cells; Tumor necrosis factor(TNF)-α; Cytokine
MeSH Terms: conditions — Wounds and Injuries; Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple-trauma patients: The patients who are diagnosed with multiple-trauma and have blood test in an emergency room. The patients with multiple-trauma are defined as the patients who have trauma in more than two regions.
  Interventions: Procedure: Multiple-trauma patients

INTERVENTIONS:
Procedure: Multiple-trauma patients — The blood samples of the patients who agreed on this research are obtained in order to check their inflammatory response factor, and then their medical records are checked to find their initial ABGA result, lactate, C-reactive protein(CRP) known as initial inflammatory response, and procalcitonin.
  A patient's whole blood is collected in the tube with ethylene diaminetetracetic acid (EDTA) treatment. A modified method of Boyum's technique is applied so as to separate polymorphonuclear neutrophils. The separated polymorphonuclear neutrophils is collected so as to check apoptosis. And then, in the separated plasma, interleukin(IL)-6 and tumor necrosis factor(TNF)-α are measured, and its correlation with oxygen saturation will be analyzed.

SUMMARY:
This study tries to find how hypoxia and hyperoxia, among types of the respiratory failure induced cell damage that can arise in the course of traumatic damage and treatment, influences apoptosis of PMN cells and IL-6 and tumor necrosis factor(TNF)-α as inflammatory cytokines.

DETAILED DESCRIPTION:
Many patients visit an emergency room because of their trauma. Trauma patients account for around 25-35% in an emergency room. Trauma is the biggest cause of acquired disabilities, and is greatly related to death and disabilities of those aged less than 44. As such, since trauma leads to lowering personal life quality and greatly influences social and economic aspects, it is greatly dealt with in public medical service.

Primarily, patients with trauma experience a lot of bleeding and respiratory failure induced by multiple causes, and furthermore is likely to have hypovolaemic shock. Secondarily, the low blood flow induced by trauma and hypovolaemic shock triggers hypoxia and systemic inflammatory response syndrome(SIRS), and therefore lowering immunity leads to compensatory anti-inflammatory response syndrome(CARS). After that, failures to keep homeostasis, such as immune dysregulation induced acute respiratory distress syndrome (ARDS), multiple organ failure(MOF), immune function reduction, and inflammation overexpression, and other additional causes damage the patients who can end up being dead without recovery.

A trauma patient is able to be exposed to multiple complications of trauma and continue to have hypoxia and hyperoxia with multiple causes in the treatment step. Hypoxia triggers multiple organ failure by cell death and lack of oxygen, and especially is sensitive to nerve cells. Hyperoxia causes the problem of immunity system stimulation by oxygen radical and hydrogen peroxide(H2O2) secretion. As such, an oxygen condition can influence organ failure and inflammatory response in various ways. These hypoxia and hyperoxia are considered to be influential on post-trauma inflammation and on Polymorphonuclear Cells(PMN) and cytokine. A patient's oxygen condition control is the basic treatment of a trauma patient and is able to influence not only the maintenance of oxygen concentration in the body, but the immunity system for keeping body homeostasis to respond to trauma.

Therefore, it is important to know how a patient's oxygen condition influences cells in order to treat the patient. Nevertheless, there is no research on how hypoxia and hyperoxia influence PMN cell and inflammatory cytokine as inflammatory cells playing a critical role in post-trauma immunity function. Therefore, this study tries to find how hypoxia and hyperoxia, among types of the respiratory failure induced cell damage that can arise in the course of traumatic damage and treatment, influences apoptosis of PMN cells and IL-6 and tumor necrosis factor(TNF)-α as inflammatory cytokines. This study is expected to be used as a fundamental material for treating relevant patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged more than 19
* The patients who are diagnosed with multiple-trauma and have blood test in an emergency room. The patients with multiple-trauma are defined as the patients who have trauma in more than two regions.

Exclusion Criteria:

* The case where the check result of blood collection and oxygen saturation is able to influence treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of this study are patients with multiple severe trauma who have visited an emergency room in one year. this study is comparative observation research and have no intervention with treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Measure interleukin(IL)-6 | At the occurrence of the event during visiting an emergency room, up to 3 hours
  * Measure in the separated plasma
  * Analyze correlation with oxygen saturation

SECONDARY OUTCOMES:
Apoptosis of PMN check | At the occurrence of the event during visiting an emergency room, up to 3 hours
  A patient's whole blood is collected in the tube with ethylene
tumor necrosis factor(TNF)-α | At the occurrence of the event during visiting an emergency room, up to 3 hours
  Measure in the separated plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Youn Kim, MD, Ph.D., Principal Investigator — Assistant Professor
Locations (1):
- Korea University Guro Hospital, Seoul, Guro-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moon S, Lee SH, Ryoo HW, Kim JK, Ahn JY, Kim SJ, Jeon JC, Lee KW, Sung AJ, Kim YJ, Lee DR, Do BS, Park SR, Lee JS. Preventable trauma death rate in Daegu, South Korea. Clin Exp Emerg Med. 2015 Dec 28;2(4):236-243. doi: 10.15441/ceem.15.085. eCollection 2015 Dec. PMID 27752603
- [Background] Deitch EA. Multiple organ failure. Pathophysiology and potential future therapy. Ann Surg. 1992 Aug;216(2):117-34. doi: 10.1097/00000658-199208000-00002. PMID 1503516
- [Background] Gillani S, Cao J, Suzuki T, Hak DJ. The effect of ischemia reperfusion injury on skeletal muscle. Injury. 2012 Jun;43(6):670-5. doi: 10.1016/j.injury.2011.03.008. Epub 2011 Apr 9. PMID 21481870
- [Background] Roumen RM, Redl H, Schlag G, Zilow G, Sandtner W, Koller W, Hendriks T, Goris RJ. Inflammatory mediators in relation to the development of multiple organ failure in patients after severe blunt trauma. Crit Care Med. 1995 Mar;23(3):474-80. doi: 10.1097/00003246-199503000-00010. PMID 7874897
- [Background] Giannoudis PV, Hildebrand F, Pape HC. Inflammatory serum markers in patients with multiple trauma. Can they predict outcome? J Bone Joint Surg Br. 2004 Apr;86(3):313-23. doi: 10.1302/0301-620x.86b3.15035. No abstract available. PMID 15125116
- [Background] Brach MA, deVos S, Gruss HJ, Herrmann F. Prolongation of survival of human polymorphonuclear neutrophils by granulocyte-macrophage colony-stimulating factor is caused by inhibition of programmed cell death. Blood. 1992 Dec 1;80(11):2920-4. PMID 1280481
- [Background] Ciesla DJ, Moore EE, Zallen G, Biffl WL, Silliman CC. Hypertonic saline attenuation of polymorphonuclear neutrophil cytotoxicity: timing is everything. J Trauma. 2000 Mar;48(3):388-95. doi: 10.1097/00005373-200003000-00004. PMID 10744274
- [Background] Elbim C, Estaquier J. Cytokines modulate neutrophil death. Eur Cytokine Netw. 2010 Mar;21(1):1-6. doi: 10.1684/ecn.2009.0183. PMID 20146984
- [Background] Greenberg S, Grinstein S. Phagocytosis and innate immunity. Curr Opin Immunol. 2002 Feb;14(1):136-45. doi: 10.1016/s0952-7915(01)00309-0. PMID 11790544
- [Background] Hsieh SC, Huang MH, Tsai CY, Tsai YY, Tsai ST, Sun KH, Yu HS, Han SH, Yu CL. The expression of genes modulating programmed cell death in normal human polymorphonuclear neutrophils. Biochem Biophys Res Commun. 1997 Apr 28;233(3):700-6. doi: 10.1006/bbrc.1997.6529. PMID 9168918
- [Background] Kim JY, Hong YS, Choi SH, Yoon YH, Moon SW, Lee SW. Effect of hypertonic saline on apoptosis of polymorphonuclear cells. J Surg Res. 2012 Nov;178(1):401-8. doi: 10.1016/j.jss.2012.01.055. Epub 2012 Mar 23. PMID 22475352
- [Background] Koller M, Clasbrummel B, Kollig E, Hahn MP, Muhr G. Major injury induces increased production of interleukin-10 in human granulocyte fractions. Langenbecks Arch Surg. 1998 Dec;383(6):460-5. doi: 10.1007/s004230050161. PMID 9921948
- [Background] Menger MD, Vollmar B. Surgical trauma: hyperinflammation versus immunosuppression? Langenbecks Arch Surg. 2004 Nov;389(6):475-84. doi: 10.1007/s00423-004-0472-0. Epub 2004 May 28. PMID 15173946
- [Background] Martin C, Boisson C, Haccoun M, Thomachot L, Mege JL. Patterns of cytokine evolution (tumor necrosis factor-alpha and interleukin-6) after septic shock, hemorrhagic shock, and severe trauma. Crit Care Med. 1997 Nov;25(11):1813-9. doi: 10.1097/00003246-199711000-00018. PMID 9366763